CLINICAL TRIAL: NCT02344576
Title: A Multicenter Trial of a Shared Decision Support Intervention for Patients and Their Caregivers Offered Destination Therapy for End-Stage Heart Failure
Brief Title: PCORI-1310-06998 Trial of a Decision Support Intervention for Patients and Caregivers Offered Destination Therapy Heart Assist Device
Acronym: DECIDE-LVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-2102; CDR-1310-06998 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; Heart-assist Devices
Keywords: heart failure; heart-assist devices; decision making; decision support techniques; hospice care; palliative care; caregivers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: Usual Care (No Intervention): Patients and caregivers will receive the current usual education and consent process for DT LVAD at each hospital. This often means viewing consent forms and industry materials.
- DT LVAD Decision Support Intervention (Experimental): In the intervention phase of the study, patients and caregivers will receive the new decision support intervention, which consists primarily of decision aid materials about DT LVAD. The standard consent process will also still take place, but will be supplemented with additional decision support.
  Interventions: Behavioral: DT LVAD Decision Support Intervention

INTERVENTIONS:
Behavioral: DT LVAD Decision Support Intervention — Decision coaching and training of staff prior to intervention, to allow for additional decision support to patients and caregivers considering DT LVAD. Decision aid materials will be used with patients and caregivers.
  Arms: DT LVAD Decision Support Intervention

SUMMARY:
The left ventricular assist device (LVAD) is growing rapidly among people dying from end-stage heart failure who are unable to get a heart transplant. These patients elect to live out the remainder of their lives dependent on a partial artificial heart-so-called destination therapy (DT). Although patients may live longer with a DT LVAD, it poses many risks, including stroke, serious infection, and bleeding. Most of these patients have other medical problems that are not fixed by the DT LVAD. Patients must be connected to electricity at all times. A caregiver is required, which often places stress on loved ones. Therefore, the decision whether or not to get a DT LVAD is often an extremely difficult one. Unfortunately, our research shows problems with the way this medical decision is currently being made in hospitals across the United States. Hospitals that offer DT LVAD treatment do not follow a standard process. The forms, pamphlets, websites, and videos used to help patients and families are biased and too difficult for most people to understand. Lastly, this is an emotional and even scary decision for most patients and their families, but the process does not help them deal with these feelings.

Using feedback from patients, caregivers, clinicians, the study team made a paper and video decision aid to help people who are offered DT LVAD make this most difficult of decisions. Unlike the information that is now available, our decision aid focuses on options, fears, and the needs of caregivers, is balanced, and is paired with training for doctors and nurses on how to best talk about DT LVAD. The investigators now propose to test the effectiveness and implementation of this intervention. The investigators will apply the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) evaluative framework to a stepped-wedge, cluster-randomized, controlled trial across 6 medical centers.

Aim 1. Evaluate the Reach and Effectiveness of the DT LVAD shared decision support intervention to improve patient and caregiver experiences.

Hypothesis 1a: The intervention will reach 90% of eligible patients. Hypothesis 1b: Post-implementation, patients and caregivers will have improved decision quality (greater knowledge and higher value-treatment concordance).

Aim 2. Assess the Adoption, Implementation, and Maintenance of the DT LVAD shared decision support intervention across multiple providers and settings.

Hypothesis 2: The intervention will be: adopted by key personnel; implemented consistently; and maintained after trial completion.

DETAILED DESCRIPTION:
The investigators plan to test the effectiveness and implementation of a shared decision support intervention for DT LVAD. Six DT LVAD programs from across the U.S. will participate in a stepped-wedge randomized study design. In this design, each site participates in both the control and intervention phase with the timing of the transition randomly assigned. Sites all begin in the control phase, where usual care consists of the current education, decision making, and informed consent process. When sites reach their randomly assigned time to transition to the intervention, their coordinators and key staff will participate in communication training and decision coaching. The pamphlet and video decision aid will be formally integrated into the existing education, decision making, and informed consent process. In both pre- and post-phases, the investigators will enroll patients and caregivers and survey them prior to their DT LVAD decision (baseline) and then at 1 month and 6 months after to determine the interventions effect on decision quality and a host of secondary outcomes. These patient- and caregiver-centered outcomes will be compared within each hospital before and after implementation to determine the effectiveness of the intervention. The investigators will also survey clinicians before, during, and after implementation of the shared decision support intervention. The implementation will be guided using the well-known RE-AIM evaluative framework (Reach, Effectiveness, Adoption, Implementation, Maintenance). Formal study of the implementation will promote widespread dissemination of this DT LVAD shared decision support.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have advanced heart failure and are being evaluated for DT LVAD
* Caregivers of patients who are being evaluated for DT LVAD

Exclusion Criteria:

* Under 18 years of age
* Non-English Speaking
* Unable to consent
* Prisoner
* Already implanted with DT LVAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Allen, MD, MHS, Principal Investigator — University of Colorado School of Medicine
Locations (6):
- United States (6):
  - University of Colorado School of Medicine, Aurora, Colorado
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine in St.Louis, St Louis, Missouri
  - Duke University Medicine, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Background] Miller LW, Guglin M. Patient selection for ventricular assist devices: a moving target. J Am Coll Cardiol. 2013 Mar 26;61(12):1209-21. doi: 10.1016/j.jacc.2012.08.1029. Epub 2013 Jan 2. PMID 23290542
- [Background] Hershberger RE, Nauman D, Walker TL, Dutton D, Burgess D. Care processes and clinical outcomes of continuous outpatient support with inotropes (COSI) in patients with refractory endstage heart failure. J Card Fail. 2003 Jun;9(3):180-7. doi: 10.1054/jcaf.2003.24. PMID 12815567
- [Background] Rose EA, Gelijns AC, Moskowitz AJ, Heitjan DF, Stevenson LW, Dembitsky W, Long JW, Ascheim DD, Tierney AR, Levitan RG, Watson JT, Meier P, Ronan NS, Shapiro PA, Lazar RM, Miller LW, Gupta L, Frazier OH, Desvigne-Nickens P, Oz MC, Poirier VL; Randomized Evaluation of Mechanical Assistance for the Treatment of Congestive Heart Failure (REMATCH) Study Group. Long-term use of a left ventricular assist device for end-stage heart failure. N Engl J Med. 2001 Nov 15;345(20):1435-43. doi: 10.1056/NEJMoa012175. PMID 11794191
- [Background] Rogers JG, Butler J, Lansman SL, Gass A, Portner PM, Pasque MK, Pierson RN 3rd; INTrEPID Investigators. Chronic mechanical circulatory support for inotrope-dependent heart failure patients who are not transplant candidates: results of the INTrEPID Trial. J Am Coll Cardiol. 2007 Aug 21;50(8):741-7. doi: 10.1016/j.jacc.2007.03.063. Epub 2007 Aug 6. PMID 17707178
- [Background] Slaughter MS, Rogers JG, Milano CA, Russell SD, Conte JV, Feldman D, Sun B, Tatooles AJ, Delgado RM 3rd, Long JW, Wozniak TC, Ghumman W, Farrar DJ, Frazier OH; HeartMate II Investigators. Advanced heart failure treated with continuous-flow left ventricular assist device. N Engl J Med. 2009 Dec 3;361(23):2241-51. doi: 10.1056/NEJMoa0909938. Epub 2009 Nov 17. PMID 19920051
- [Background] Grady KL, Meyer PM, Dressler D, Mattea A, Chillcott S, Loo A, White-Williams C, Todd B, Ormaza S, Kaan A, Costanzo MR, Piccione W. Longitudinal change in quality of life and impact on survival after left ventricular assist device implantation. Ann Thorac Surg. 2004 Apr;77(4):1321-7. doi: 10.1016/j.athoracsur.2003.09.089. PMID 15063260
- [Background] McIlvennan CK, Magid KH, Ambardekar AV, Thompson JS, Matlock DD, Allen LA. Clinical outcomes after continuous-flow left ventricular assist device: a systematic review. Circ Heart Fail. 2014 Nov;7(6):1003-13. doi: 10.1161/CIRCHEARTFAILURE.114.001391. Epub 2014 Oct 7. PMID 25294625
- [Background] Kirklin JK, Naftel DC, Kormos RL, Stevenson LW, Pagani FD, Miller MA, Baldwin JT, Young JB. Fifth INTERMACS annual report: risk factor analysis from more than 6,000 mechanical circulatory support patients. J Heart Lung Transplant. 2013 Feb;32(2):141-56. doi: 10.1016/j.healun.2012.12.004. PMID 23352390
- [Background] Flint KM, Matlock DD, Lindenfeld J, Allen LA. Frailty and the selection of patients for destination therapy left ventricular assist device. Circ Heart Fail. 2012 Mar 1;5(2):286-93. doi: 10.1161/CIRCHEARTFAILURE.111.963215. No abstract available. PMID 22438521
- [Background] Allen LA, Stevenson LW, Grady KL, Goldstein NE, Matlock DD, Arnold RM, Cook NR, Felker GM, Francis GS, Hauptman PJ, Havranek EP, Krumholz HM, Mancini D, Riegel B, Spertus JA; American Heart Association; Council on Quality of Care and Outcomes Research; Council on Cardiovascular Nursing; Council on Clinical Cardiology; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Surgery and Anesthesia. Decision making in advanced heart failure: a scientific statement from the American Heart Association. Circulation. 2012 Apr 17;125(15):1928-52. doi: 10.1161/CIR.0b013e31824f2173. Epub 2012 Mar 5. No abstract available. PMID 22392529
- [Background] McIlvennan CK, Allen LA. To DT or not to DT, that is the question: working toward a comprehensive, patient-centered perspective on left ventricular assist device for destination therapy. Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):13-4. doi: 10.1161/CIRCOUTCOMES.113.000762. Epub 2014 Jan 14. No abstract available. PMID 24425698
- [Background] Baker K, Flattery M, Salyer J, Haugh KH, Maltby M. Caregiving for patients requiring left ventricular assistance device support. Heart Lung. 2010 May-Jun;39(3):196-200. doi: 10.1016/j.hrtlng.2009.07.007. Epub 2009 Oct 1. PMID 20457339
- [Background] Fowler FJ Jr, Levin CA, Sepucha KR. Informing and involving patients to improve the quality of medical decisions. Health Aff (Millwood). 2011 Apr;30(4):699-706. doi: 10.1377/hlthaff.2011.0003. PMID 21471491
- [Background] McIlvennan CK, Allen LA, Nowels C, Brieke A, Cleveland JC, Matlock DD. Decision making for destination therapy left ventricular assist devices: "there was no choice" versus "I thought about it an awful lot". Circ Cardiovasc Qual Outcomes. 2014 May;7(3):374-80. doi: 10.1161/CIRCOUTCOMES.113.000729. Epub 2014 May 13. PMID 24823949
- [Background] O'Connor AM, Wennberg JE, Legare F, Llewellyn-Thomas HA, Moulton BW, Sepucha KR, Sodano AG, King JS. Toward the 'tipping point': decision aids and informed patient choice. Health Aff (Millwood). 2007 May-Jun;26(3):716-25. doi: 10.1377/hlthaff.26.3.716. PMID 17485749
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Iacovetto MC, Matlock DD, McIlvennan CK, Thompson JS, Bradley W, LaRue SJ, Allen LA. Educational resources for patients considering a left ventricular assist device: a cross-sectional review of internet, print, and multimedia materials. Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):905-11. doi: 10.1161/CIRCOUTCOMES.114.000892. Epub 2014 Oct 14. PMID 25316772
- [Background] Coulter A, Stilwell D, Kryworuchko J, Mullen PD, Ng CJ, van der Weijden T. A systematic development process for patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S2. doi: 10.1186/1472-6947-13-S2-S2. Epub 2013 Nov 29. PMID 24625093
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Matlock DD, Spatz ES. Design and testing of tools for shared decision making. Circ Cardiovasc Qual Outcomes. 2014 May;7(3):487-92. doi: 10.1161/CIRCOUTCOMES.113.000289. Epub 2014 Apr 8. No abstract available. PMID 24714602
- [Background] Volandes AE, Ariza M, Abbo ED, Paasche-Orlow M. Overcoming educational barriers for advance care planning in Latinos with video images. J Palliat Med. 2008 Jun;11(5):700-6. doi: 10.1089/jpm.2007.0172. PMID 18588401
- [Background] Mdege ND, Man MS, Taylor Nee Brown CA, Torgerson DJ. Systematic review of stepped wedge cluster randomized trials shows that design is particularly used to evaluate interventions during routine implementation. J Clin Epidemiol. 2011 Sep;64(9):936-48. doi: 10.1016/j.jclinepi.2010.12.003. Epub 2011 Mar 16. PMID 21411284
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. Health Educ Res. 2006 Oct;21(5):688-94. doi: 10.1093/her/cyl081. Epub 2006 Aug 31. PMID 16945984
- [Background] Sepucha KR, Levin CA, Uzogara EE, Barry MJ, O'Connor AM, Mulley AG. Developing instruments to measure the quality of decisions: early results for a set of symptom-driven decisions. Patient Educ Couns. 2008 Dec;73(3):504-10. doi: 10.1016/j.pec.2008.07.009. Epub 2008 Aug 20. PMID 18718734
- [Background] Helfrich CD, Li YF, Sharp ND, Sales AE. Organizational readiness to change assessment (ORCA): development of an instrument based on the Promoting Action on Research in Health Services (PARIHS) framework. Implement Sci. 2009 Jul 14;4:38. doi: 10.1186/1748-5908-4-38. PMID 19594942
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Heyland DK, Cook DJ, Rocker GM, Dodek PM, Kutsogiannis DJ, Skrobik Y, Jiang X, Day AG, Cohen SR; Canadian Researchers at the End of Life Network. The development and validation of a novel questionnaire to measure patient and family satisfaction with end-of-life care: the Canadian Health Care Evaluation Project (CANHELP) Questionnaire. Palliat Med. 2010 Oct;24(7):682-95. doi: 10.1177/0269216310373168. Epub 2010 Jul 6. PMID 20605850
- [Derived] Raymer DS, Allen LA, Chaussee EL, McIlvennan CK, Thompson JS, Fairclough DL, Dunlay SM, Matlock DD, Larue SJ. Health Literacy in Patients Considering a Left Ventricular Assist Device: Findings From the DECIDE-LVAD Trial. J Card Fail. 2022 Aug;28(8):1318-1325. doi: 10.1016/j.cardfail.2022.04.009. Epub 2022 May 13. PMID 35569806
- [Derived] McIlvennan CK, Jones J, Makic M, Meek PM, Chaussee E, Thompson JS, Matlock DD, Allen LA. Stress and Coping Among Family Caregivers of Patients With a Destination Therapy Left Ventricular Assist Device: A Multicenter Mixed Methods Study. Circ Heart Fail. 2021 Oct;14(10):e008243. doi: 10.1161/CIRCHEARTFAILURE.120.008243. Epub 2021 Sep 1. PMID 34465131
- [Derived] Knoepke CE, Chaussee EL, Matlock DD, Thompson JS, McIlvennan CK, Ambardekar AV, Schaffer EM, Khazanie P, Scherer L, Arnold RM, Allen LA. Changes over Time in Patient Stated Values and Treatment Preferences Regarding Aggressive Therapies: Insights from the DECIDE-LVAD Trial. Med Decis Making. 2022 Apr;42(3):404-414. doi: 10.1177/0272989X211028234. Epub 2021 Jul 23. PMID 34296623
- [Derived] Matlock DD, McIlvennan CK, Thompson JS, Morris MA, Venechuk G, Dunlay SM, LaRue SJ, Lewis EF, Patel CB, Blue L, Chaussee EL, Glasgow RE, Walsh MN, Allen LA. Decision Aid Implementation among Left Ventricular Assist Device Programs Participating in the DECIDE-LVAD Stepped-Wedge Trial. Med Decis Making. 2020 Apr;40(3):289-301. doi: 10.1177/0272989X20915227. PMID 32428430
- [Derived] McIlvennan CK, Matlock DD, Allen LA, Thompson JS, Ranby KW, Sannes TS. Perceived Stress and Depressive Symptoms as Predictors of Decisional Conflict in Dyads Considering a Left Ventricular Assist Device. Circ Cardiovasc Qual Outcomes. 2020 Mar;13(3):e006155. doi: 10.1161/CIRCOUTCOMES.119.006155. Epub 2020 Mar 9. PMID 32148099
- [Derived] Warraich HJ, Allen LA, Blue LJ, Chaussee EL, Thompson JS, McIlvennan CK, Flint KM, Matlock DD, Patel CB. Comorbidities and the decision to undergo or forego destination therapy left ventricular assist device implantation: An analysis from the Trial of a Shared Decision Support Intervention for Patients and their Caregivers Offered Destination Therapy for End-Stage Heart Failure (DECIDE-LVAD) study. Am Heart J. 2019 Jul;213:91-96. doi: 10.1016/j.ahj.2019.04.008. Epub 2019 Apr 25. PMID 31129442
- [Derived] McIlvennan CK, Matlock DD, Thompson JS, Dunlay SM, Blue L, LaRue SJ, Lewis EF, Patel CB, Fairclough DL, Leister EC, Swetz KM, Baldridge V, Walsh MN, Allen LA. Caregivers of Patients Considering a Destination Therapy Left Ventricular Assist Device and a Shared Decision-Making Intervention: The DECIDE-LVAD Trial. JACC Heart Fail. 2018 Nov;6(11):904-913. doi: 10.1016/j.jchf.2018.06.019. Epub 2018 Oct 10. PMID 30316931
- [Derived] Allen LA, McIlvennan CK, Thompson JS, Dunlay SM, LaRue SJ, Lewis EF, Patel CB, Blue L, Fairclough DL, Leister EC, Glasgow RE, Cleveland JC Jr, Phillips C, Baldridge V, Walsh MN, Matlock DD. Effectiveness of an Intervention Supporting Shared Decision Making for Destination Therapy Left Ventricular Assist Device: The DECIDE-LVAD Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):520-529. doi: 10.1001/jamainternmed.2017.8713. PMID 29482225
- [Derived] McIlvennan CK, Thompson JS, Matlock DD, Cleveland JC Jr, Dunlay SM, LaRue SJ, Lewis EF, Patel CB, Walsh MN, Allen LA. A Multicenter Trial of a Shared Decision Support Intervention for Patients and Their Caregivers Offered Destination Therapy for Advanced Heart Failure: DECIDE-LVAD: Rationale, Design, and Pilot Data. J Cardiovasc Nurs. 2016 Nov/Dec;31(6):E8-E20. doi: 10.1097/JCN.0000000000000343. PMID 27203272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Occurred from June 2015-Jan 2017 in both the inpatient and outpatient setting. Patients were identified by the study team when a destination therapy left ventricular assist device evaluation was initiated; caregivers were identified by the medical team or patient. Recruitment and data collection were identical across control and intervention arms.
Pre-assignment Details: This study had a stepped-wedge design. All 6 sites started in the control phase, and then were transitioned to the intervention phase over pre-determined and randomly assigned time points (all sites ended in intervention). Participant assignment to control or intervention was determined by phase the site was in at time of participant enrollment.
Groups:
- Patient Control: Patients being considered for destination therapy (DT) LVAD therapy enrolled during the control phase. These patients receive the usual care education and consent process for DT LVAD at each hospital. This often means viewing consent forms and industry materials.
- Patient Intervention: Patients being considered for DT LVAD therapy enrolled during the intervention phase. These patients receive the intervention, consisting of staff trained in decision making and use of a decision aid pamphlet and video during education.
- Caregiver Control: Caregivers of patients being considered for DT LVAD therapy enrolled during the control phase. These caregivers receive the usual care education and consent process for DT LVAD at each hospital. This often means viewing consent forms and industry materials.
- Caregiver Intervention: Caregivers of patients being considered for DT LVAD enrolled during the intervention phase. These caregivers receive the intervention, consisting of staff trained in decision making and use of a decision aid pamphlet and video during education.
Period: Enrollment
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Started | 142 (Includes 7 patients who agreed to medical record review only and were excluded from further analysis) | 121 (Includes 8 patients who agreed to medical record review only and were excluded from further analysis) | 111 | 71
Agreed to Survey Data Collection | 135 | 113 | 111 | 71
Completed | 135 | 113 | 111 | 71
Not Completed | 7 | 8 | 0 | 0
Not completed — Agreed to Medical Record Review Only | 7 | 8 | 0 | 0
Period: 1-Month Follow-Up
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Started | 135 | 113 | 111 | 71
Completed 1-Month Survey | 104 | 79 | 89 | 53
Completed | 117 (Includes 13 patients who were still enrolled at 1-month but did not complete the 1-month survey.) | 86 (Includes 7 patients who were still enrolled at 1-month but did not complete the 1-month survey.) | 92 (Includes 3 caregivers who were still enrolled at 1-month but did not complete the 1-month survey.) | 58 (Includes 5 caregivers who were still enrolled at 1-month but did not complete the 1-month survey.)
Not Completed | 18 | 27 | 19 | 13
Not completed — Death | 13 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 14 | 8 | 10
Not completed — Lost to Follow-up | 2 | 5 | 11 | 3
Period: 6-Month Follow-Up
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Started | 117 | 86 | 92 | 58
Completed 6-Month Survey | 98 | 67 | 78 | 50
Completed | 98 | 67 | 78 | 50
Not Completed | 19 | 19 | 14 | 8
Not completed — Death | 14 | 14 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 4 | 5 | 13 | 6
Period: 12-Month Medical Record Follow-Up
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Started (12-month period applicable to patient participants only.) | 98 | 67 | 78 (This period not applicable to caregivers, as medical record review was completed for patients only.) | 50 (This period not applicable to caregivers, as medical record review was completed for patients only.)
Completed (12-month period applicable to patient participants only.) | 98 | 67 | 78 (This period not applicable to caregivers, as medical record review was completed for patients only.) | 50 (This period not applicable to caregivers, as medical record review was completed for patients only.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics collected for patient and caregiver participants only; does not apply to the "Sites" arm. Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in baseline characteristics analysis, as this data was primarily collected in surveys.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention | Total
Number analyzed (Participants) | 135 | 113 | 111 | 71 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.7) | 63.2 (10.2) | 60.2 (11.2) | 62.2 (11.5) | 62.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 15 | 92 | 62 | 193
  Male | 111 | 98 | 19 | 9 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 2 | 9
  Not Hispanic or Latino | 124 | 100 | 108 | 64 | 396
  Unknown or Not Reported | 9 | 10 | 1 | 5 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 0 | 4
  Asian | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 12 | 14 | 6 | 51
  White | 104 | 88 | 91 | 59 | 342
  More than one race | 4 | 2 | 3 | 1 | 10
  Unknown or Not Reported | 4 | 9 | 1 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 135 | 113 | 111 | 71 | 430
Mean Cognitive Function Score [Mean (Standard Deviation); unit: scores on a scale] — Measured with the Short Portable Mental Status Questionnaire. Number of incorrect answers out of 10 questions, scale range of 0 to 10, with lower number indicating better cognitive function.
  scores on a scale | 0.7 (1.55) | 0.66 (1.25) | 0.60 (1.69) | 0.39 (1.29) | 0.61 (1.49)
Mean Literacy Score, as measured by Revised (REALM-R) measure [Mean (Standard Deviation); unit: scores on a scale] — Measured with the Rapid Estimate of Adult Literacy in Medicine, Revised (REALM-R) measure. Number of correctly read words out of 8 listed, scale range of 0-8, with higher number indicating higher literacy.
  scores on a scale | 6.93 (1.9) | 6.95 (2.0) | 7.46 (1.50) | 7.70 (0.98) | 7.24 (1.61)
Numeracy Score [Mean (Standard Deviation); unit: units on a scale] — Measured with the Subjective Numeracy Score measure. Range of 1-6, higher numeracy toward 6.
  units on a scale | 4.03 (1.10) | 4.21 (1.13) | 4.04 (1.28) | 4.31 (1.19) | 4.13 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Reach of Intervention
Description: Reach: The proportion of the target population who participate in the intervention. We will assess the percentage of patients and caregivers that receive the pamphlet and video decision aids.
Time Frame: Baseline 2 (post-education: average 3 days after enrollment)
Population: Reach pertains to only those participants in the intervention phase, and therefore the control arms are not included here.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Intervention | Caregiver Intervention
Number analyzed (Participants) | 113 | 71
Participants | 107 | 64

2. Primary Outcome: Effectiveness of Intervention: Knowledge
Description: Effectiveness: Assessed based on if the decision support intervention led to a quality decision. Decision quality is defined as "the extent to which the implemented decision reflects the considered preferences of a well-informed patient." By this definition, a decision is "a quality decision" if the treatment chosen is concordant with a knowledgeable patient's values. Decision quality measures consist of 2 domains: knowledge and values.
  This is part one of the decision quality measure:
  -Knowledge: DT LVAD knowledge score improvement from Baseline 1 (enrollment) to Baseline 2 (post-education), measured by percentage of score improvement (scale of 0-100%).
Time Frame: Baseline 1 (enrollment), Baseline 2 (post-education: average 3 days after enrollment)
Population: Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in Effectiveness analysis, as this data was collected in surveys.
Measure: Mean (Standard Error); unit: percentage of score improvement
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 135 | 113 | 111 | 71
percentage of score improvement | 5.4 (1.6) | 10.9 (1.9) | 9.1 (1.7) | 13.9 (2.2)

3. Primary Outcome: Adoption of Intervention
Description: Adoption: The absolute number of settings who are willing to initiate a program. We will assess the number of sites who agreed to be part of the study and who initiate intervention at intervention period.
Time Frame: At time of intervention phase start
Population: Adoption is measured by sites only; does not apply to the "Patient" and "Caregiver" arms. Adoption pertains to only the intervention phase; thus, for "overall number of participants analyzed", includes patients and caregivers in intervention phase only.
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Groups:
- Sites: Hospital's left ventricular assist device (LVAD) programs implementing the intervention as the new standard of care at their site. Sites start in the usual care control phase and then are randomly phased into the intervention phase over time. The intervention consists of decision coaching and communication training of staff and use of a decision aid pamphlet and video during patient and caregiver education.
Arm/Group | Sites
Number analyzed (Participants) | 184
Number analyzed (Sites) | 6
Sites | 6

4. Primary Outcome: Implementation of Intervention
Description: Implementation: The extent to which the intervention is implemented as intended. We will assess implementation by surveying the consistency of decision aid delivery by the sites to the enrolled patients.
Time Frame: Baseline 2 (post-education: average 3 days after enrollment)
Population: Implementation was collected for patient participants only; does not apply to the "Caregiver" arm. Implementation pertains to only patients in the intervention phase; control arms are not included here.Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included.
Measure: Number; unit: percentage of eligible participants
Arm/Group | Patient Intervention
Number analyzed (Participants) | 113
percentage of eligible participants
  Provided by Clinician (Non-Study Personnel) | 98.3
  Patient Kept Decision Aids | 90.9
  Clinician Went through Pamphlet with Patient | 26.4
  Patient Viewed Video in Clinical Setting | 46.8

5. Primary Outcome: Maintenance of Intervention
Description: Maintenance: Assessing whether sites decide at the conclusion of the study to maintain, modify, or discontinue a program. We will assess maintenance by counting the number of sites who continue the intervention after the study enrollment period has ended.
Time Frame: 6 months after study enrollment end date
Population: Maintenance is measured by sites only; does not apply to the "Patient" and "Caregiver" arms. Maintenance pertains to only the intervention phase; thus, for "overall number of participants analyzed", includes patients and caregivers in intervention phase only.
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Sites
Number analyzed (Participants) | 184
Number analyzed (Sites) | 6
Sites | 5

6. Secondary Outcome: Changes in Decision Conflict (Decision Conflict Scale)
Description: Decision Conflict Scale: 16-items, scoring 0-100 with higher score indicating greater decisional conflict.
Time Frame: Baseline 1 (enrollment), Baseline 2 (post-education: average 3 days after enrollment), 1 Month Follow-Up, and 6 Month Follow-Up
Population: Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in Decision Conflict analysis, as this data was collected in surveys.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 135 | 113 | 111 | 71
units on a scale
  Baseline 1 Survey Score | 20.2 (1.99) | 23.4 (2.24) | 19.0 (2.06) | 21.4 (2.59)
  Baseline 2 Survey Score | 16.5 (1.95) | 18.4 (2.23) | 9.70 (1.90) | 18.8 (2.40)
  1-Month Follow-Up Survey Score | 15.5 (1.89) | 17.9 (2.17) | 13.1 (2.09) | 19.5 (2.62)
  6-Month Follow-Up Survey Score | 15.4 (1.89) | 14.2 (2.21) | 11.9 (1.98) | 17.4 (2.52)

7. Secondary Outcome: Changes in Decision Regret (Decision Regret Scale)
Description: Decision Regret Scale: 5-items, scoring 0-100 with higher score indicating greater decision regret.
Time Frame: 1 Month Follow-Up, and 6 Month Follow-Up
Population: Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in Decision Regret analysis, as this data was collected in surveys.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 135 | 113 | 111 | 71
units on a scale
  1-Month Follow-Up Survey | 14.3 (2.15) | 17.9 (2.84) | 11.2 (2.37) | 17.5 (3.32)
  6-Month Follow-Up Survey | 12.1 (2.28) | 19.1 (2.96) | 10.4 (2.46) | 17.1 (3.38)

8. Secondary Outcome: Changes in Stress and Depression (Perceived Stress Scale; Patient Health Questionnaire-2)
Description: Perceived Stress Scale (collected at Baseline 1 and 6-month follow-up only):10-items, scoring 0-40 with higher score indicating greater stress.; Patient Health Questionnaire-2: 2-items, score of 0-6 with higher score indicating greater depression.
Time Frame: Baseline 1 (enrollment), 1 month Follow-Up, and 6 Month Follow-Up
Population: Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in Stress and Depression analysis, as this data was collected in surveys.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 135 | 113 | 111 | 71
units on a scale
  Stress: Baseline 1 Survey Score | 16.1 (0.68) | 14.1 (0.81) | 14.3 (0.86) | 16.4 (1.06)
  Stress: 6-Month Follow-Up Survey Score | 12.6 (0.82) | 11.9 (1.03) | 12.1 (1.00) | 12.7 (1.24)
  Depression: Baseline 1 Survey Score | 1.80 (0.21) | 1.56 (0.24) | 0.79 (0.22) | 1.04 (0.26)
  Depression: 1-Month Follow-Up Survey Score | 1.64 (0.23) | 1.39 (0.26) | 0.80 (0.24) | 1.35 (0.29)
  Depression: 6-Month Follow-Up Survey Score | 1.06 (0.21) | 0.97 (0.25) | 0.54 (0.21) | 0.69 (0.24)

9. Secondary Outcome: Changes in Quality of Life (EuroQol Visual Analogue Scale [Patients Only])
Description: EuroQol Visual Analogue Scale (patients only): 1-item scale, score of 0-100 with 0 being "worst imaginable health state" and 100 being "best imaginable health state".
Time Frame: Baseline 1 (enrollment), 1 month Follow-Up, and 6 month Follow-Up
Population: EuroQol Visual Analogue Scale was collected for patient participants only; does not apply to the "Caregiver" arm. Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in EuroQol Visual Analogue Scale analysis, as this data was collected in surveys.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patient Control | Patient Intervention
Number analyzed (Participants) | 135 | 113
units on a scale
  Baseline 1 Survey Score | 44.6 (2.69) | 48.6 (3.07)
  1-Month Follow-Up Survey Score | 64.3 (2.67) | 60.5 (3.13)
  6-Month Follow-Up Survey Score | 69.6 (2.57) | 68.8 (3.07)

10. Secondary Outcome: Changes in Caregiver's Preparedness for Caregiving (Preparedness for Caregiving Scale [Caregivers Only])
Description: Preparedness for Caregiving Scale (caregivers only): 8-items, scoring 0-4 with higher score indicating more preparedness.
Time Frame: Baseline 1 (enrollment), 1 month Follow-Up, and 6 month Follow-Up
Population: Preparedness for Caregiving Scale was collected for caregiver participants only; does not apply to the "Patient" arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 111 | 71
units on a scale
  Baseline 1 Survey Score | 3.05 (0.10) | 2.81 (0.13)
  1-Month Follow-Up Survey Score | 3.17 (0.10) | 3.02 (0.13)
  6-Month Follow-Up Survey Score | 3.24 (0.11) | 2.99 (0.13)

11. Secondary Outcome: Changes in Bereaved Caregiver Satisfaction With End-of-Life Care (Canadian Health Care Evaluation Project - Bereavement Questionnaire [Bereaved Caregivers Only])
Description: Canadian Health Care Evaluation Project - Bereavement Questionnaire (bereaved caregivers only): Score of 0-100 with higher score indicating greater satisfaction.
Time Frame: 6 Month Follow-Up
Population: Bereaved Caregiver Satisfaction was collected for caregiver participants only; does not apply to the "Patient" arm. This measure was also collected among bereaved caregivers only; 11 bereaved caregivers responded.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 6 | 5
units on a scale | 73.0 (6.0) | 62.0 (10.2)

12. Secondary Outcome: Changes in Preferences for Control of Medical Decisions (Control Preferences Scale [Patients Only])
Description: Control Preferences Scale (patients only) includes 2 parts: "Preferred" and "Actual" ("Actual" at 1-Month and 6-Month only). Each is a 1-item question with 5-answer options, assessing preferred or actual control in decision making. "Active role" indicated if 1 of first 3 answer options were selected: for "Preferred", those 3 answer options were "I prefer to make the final selection about which treatment I will receive", "I prefer to make the final selection of my treatment after seriously considering my doctor's opinion", or "I prefer that my doctor and I share responsibility for deciding which treatment is best"; for "Actual", answer options were "I made the final selection about which treatment I would receive", "I made the final selection of my treatment after seriously considering my doctor's opinion", or "My doctor and I shared responsibility for deciding which was treatment best for me". The percentage of patients who selected an "active" response option was calculated.
Time Frame: Baseline 1 (enrollment), 1 Month Follow-Up, and 6 Month Follow-Up
Population: Control Preferences Scale was collected for patient participants only; does not apply to the "Caregiver" arm. Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in Control Preferences Scale analysis, as this data was collected in surveys.
Measure: Number; unit: percentage of patients in active role
Arm/Group | Patient Control | Patient Intervention
Number analyzed (Participants) | 135 | 113
percentage of patients in active role
  Preferred: Baseline 1 Survey Score | 84.1 | 83.6
  Preferred: 1-Month Follow-Up Survey Score | 86.6 | 89.8
  Preferred: 6-Month Follow-Up Survey Score | 86.7 | 92.4
  Actual: 1-Month Follow-Up Survey Score | 87.5 | 83.6
  Actual: 6-Month Follow-Up Survey Score | 85.8 | 89.4

13. Secondary Outcome: Changes in Illness Acceptance (PEACE Illness Acceptance Measure (Patients Only)
Description: PEACE Illness Acceptance Measure (patients only): 2 part measure: part 1 measures illness acceptances (questions 1-5 of 12-items), scoring 5-20 with higher score indicating greater acceptance of illness; part 2 measures struggle with illness (questions 6-12 of 12-items), scoring 7-28 with higher score indicating greater struggle with illness.
Time Frame: Baseline 1 (enrollment), 1 Month Follow-Up, and 6 Month Follow-Up
Population: PEACE Illness Acceptance Measure was collected for patient participants only; does not apply to the "Caregiver" arm. Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in PEACE Measure analysis, as this data was collected in surveys.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patient Control | Patient Intervention
Number analyzed (Participants) | 135 | 113
units on a scale
  Acceptance of Illness: Baseline 1 Survey Score | 17.5 (0.26) | 17.1 (0.31)
  Acceptance of Illness: 1-Month Survey Score | 17.4 (0.27) | 17.4 (0.32)
  Acceptance of Illness: 6-Month Survey Score | 17.5 (0.28) | 18.2 (0.34)
  Struggle with Illness: Baseline 1 Survey Score | 14.0 (0.42) | 13.1 (0.50)
  Struggle with Illness: 1-Month Survey Score | 13.6 (0.47) | 12.9 (0.57)
  Struggle with Illness: 6-Month Survey Score | 12.9 (0.50) | 12.0 (0.62)

14. Secondary Outcome: Changes in Family Satisfaction With Patient's Care (Family Satisfaction With Care [Caregivers Only])
Description: Family Satisfaction with Care (caregivers only): The 10-item "Family Satisfaction with Decision-Making around Care of Critically Ill Patients" subscale of the Family Satisfaction with Care in the Intensive Care Unit-24. Scoring for each question was on a scale of 0-100, with 0 indicating low satisfaction and 100 indicating high satisfaction; combined total of all 10 questions was taken for final mean score of 0-100 (higher score indicating higher satisfaction).
Time Frame: 1 Month Follow-Up, and 6 Month Follow-Up
Population: Family Satisfaction with Care was collected for caregiver participants only; does not apply to the "Patient" arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 111 | 71
units on a scale
  1-Month Follow-Up Survey | 76.2 (1.93) | 74.8 (2.63)
  6-Month Follow-Up Survey | 74.5 (2.11) | 77.0 (2.81)

15. Secondary Outcome: Changes in Patient Treatment Status (Medical Record Review (Patients Only)
Description: Medical record review (patients only): Treatment received by 6 months, below numbers reported as number of participants who received an LVAD.
Time Frame: 6 Month Follow-Up
Population: Medical record data was collected for patient participants only; does not apply to the "Caregiver" arm. Those patients who agreed to medical record review only (n=7 control, n=8 intervention) were not included in medical record data analysis, as this data was collected in surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Control | Patient Intervention
Number analyzed (Participants) | 135 | 113
Participants | 110 | 54

16. Primary Outcome: Effectiveness of Intervention: Values-Choice Concordance
Description: Effectiveness: Assessed based on if the decision support intervention led to a quality decision (see "Knowledge" outcome measure for full description). This is part two of the decision quality measure:
  -Values: Concordance between patients' and caregivers' stated values and their treatment choice at 1-Month. Values measured on a Likert scale of 1-10, with 1 being "Do everything I can to live longer, even if that means having major surgery and being dependent on a machine" and 10 being "Live with whatever time I have left, without going through major surgery or being dependent on a machine"; correlated with patient-reported treatment decision of accepted or declined DT LVAD. Measured by kendall's tau correlation coefficient, which ranges 1 to -1, score closer to 1 or -1 shows greater values-choice concordance (a correlation coefficient of 0 means no concordance). Confidence intervals obtained from the distribution after 500 bootstrap samples (2.5, 97.5 percentiles).
Time Frame: Baseline 1 (enrollment) and 1 Month Follow-Up
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: kendall's tau correlation coefficient
Arm/Group | Patient Control | Patient Intervention | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 135 | 113 | 111 | 71
kendall's tau correlation coefficient | 0.17 [0.15 to 0.29] | 0.48 [0.28 to 0.63] | 0.12 [-0.17 to 0.34] | 0.49 [0.26 to 0.67]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 1-Month, 6-Month and 12-Month follow-up, reported here cumulatively.
Description: Medical adverse events reported for patient participants only, therefore the caregiver arms are not included. This study's aims focus on patients' medical history/treatment/outcomes only. Thus, caregiver medical record data was not collected (caregiver medical data is not relevant for outcomes). Survey outcomes data solely were collected for caregivers. Medical data were collected for patients only; thus, adverse events include the patient arms only.
Arm/Group | Patient Control | Patient Intervention
All-Cause Mortality (participants affected / at risk) | 31/135 | 39/113
Serious Adverse Events (participants affected / at risk) | 87/135 | 57/113
Other Adverse Events (participants affected / at risk) | 117/135 | 78/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Control (N=135) | Patient Intervention (N=113)
Neurological Event (Cardiac disorders) | 18 | 17
Major Bleeding Event (Blood and lymphatic system disorders) | 64 | 38
Right Ventricular Assist Device Implant (Cardiac disorders) | 4 | 2
Major Infection (Infections and infestations) | 56 | 26
Endotrachael Mechanical Ventilation (Cardiac disorders) | 36 | 26 — Need for endotrachael mechanical ventilation other than for the 72 hours around LVAD implant surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Control (N=135) | Patient Intervention (N=113)
Inotrope Support (Cardiac disorders) | 107 | 73
Renal Replacement Therapy/Dialysis (Renal and urinary disorders) | 17 | 8
Implantable Cardioverter Defibrillator Shocks (Cardiac disorders) | 26 | 12
Psychiatric Episode (Psychiatric disorders) | 16 | 11

LIMITATIONS AND CAVEATS:
Limitations include: 1) Missing data were somewhat frequent and concentrated among the group of patients who did not undergo implantation of DT LVAD. Our models adjusted for missing data as possible. 2) The population was mostly white males.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02344576/Prot_000.pdf
  • Informed Consent Form (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02344576/ICF_001.pdf
  • Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02344576/SAP_002.pdf